CLINICAL TRIAL: NCT00444314
Title: Phase II Study of 2-Methoxyestradiol Nanocrystal Colloidal Dispersion Alone and in Combination With Sunitinib Malate in Patients With Metastatic Renal Cell Carcinoma Progressing on Sunitinib Malate
Brief Title: Phase 2 Study of Panzem® NCD Alone and Combined With Sunitinib Malate in Patients With Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Chief Medical Officer, EntreMed, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ME-CLN-008
Record Dates: First submitted 2007-03-06; First posted 2007-03-07 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-08

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

ARMS (2):
- A (Experimental)
  Interventions: Drug: Panzem® NCD
- B (Experimental)
  Interventions: Drug: Panzem® NCD; Drug: Sunitinib Malate

INTERVENTIONS:
Drug: Panzem® NCD — NCD suspension, 1500 mg TID daily for 6 week cycles
Drug: Sunitinib Malate — Sunitinib Malate, highest tolerated dose (patient's current dose), daily oral administration for 4 weeks, with 2 week break in 6 week cycle
  Other Names: Sutent
  Arms: B

SUMMARY:
This open-label, multicenter, Phase 2 trial, will assess the anti tumor activity, safety and pharmacodynamics, of Panzem® NCD with or without Sunitinib Malate in patients with metastatic renal cell carcinoma progressing on Sunitinib Malate.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically confirmed renal cell cancer with a component of clear cell carcinoma and evidence of metastasis (pure sarcomatoid variant cancers and collecting duct malignancies will be excluded).
2. Patients must have measurable disease, defined as at least one target lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to 2 times the slice width with spiral CT scan (i.e. 10 mm if the CT slice width is 5 mm, 14 mm if the CT slice width is 7 mm).
3. Patients must have previously received or be currently receiving sunitinib malate (Sutent) with evidence of disease progression while receiving sunitinib malate (as evident by new lesions on CT/MRI/bone scan or unequivocal growth in measurable tumor lesions).

   Note: Patients will be stratified to:

   A: Patients previously treated with sunitinib malate. At least 4 week washout since last treatment administered is required before patient is eligible for study. Once patients meet all other eligibility criteria, they will be treated with Panzem® NCD alone.

   B: Patients currently still on sunitinib. Patients will continue to receive their current dose/schedule of sunitinib. Once eligibility determined, patients will be started on Panzem® NCD concurrently with their sunitinib. No drug washout of sunitinib malate is required for this stratification.

   Note: Enrollment to the individual stratification will stop once that stratification has met its accrual goal.
4. Age greater than or equal to 18 years.
5. Life expectancy of greater than 3 months.
6. ECOG performance status 0-2 (see Appendix A).
7. Patients must have normal organ and marrow function as defined below:

   * leukocytes greater than or equal to 3,000/μL
   * absolute neutrophil count greater than or equal to 1,200/μL
   * hemoglobin greater than or equal to 9.0 g/dl (patient may be transfused to this level)
   * platelets greater than or equal to 100,000/μL
   * total bilirubin within normal institutional limits
   * AST(SGOT)/ALT(SGPT)less than or equal to 2.5 X institutional upper limit of normal
   * creatinine less than or equal to 1.5 x institutional upper limit of normal
8. Adequate cardiac function by history. If the patient has any history of cardiac disease (prior myocardial infarction, congestive heart failure, etc.), a normal echocardiogram or multigated acquisition (MUGA) scan will be required (LVEF greater than or equal to institutional lower limit of normal).
9. No evidence for uncontrolled hypertension as documented by 2 baseline blood pressure readings taken at least 1 hour apart. The systolic blood pressure must be less than or equal to 140 mmHg and the diastolic blood pressure less than or equal to 90 mmHg. Patients are allowed to be on anti-hypertensive medications.
10. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. No major surgery, radiotherapy, chemotherapy, cytokine therapy or other experimental therapy is permitted within 4 weeks of treatment initiation. Patients must recover to baseline or grade 1 from any clinically significant adverse event experienced during those prior therapies.
2. Patients may not be concurrently receiving any other investigational agents while participating on this study.
3. Patients with active brain metastases are excluded. Previously treated brain metastasis will be allowed provided that the patient is clinically stable (off systemic steroids and not on antiepileptic agents) with a repeat imaging study (within 4 weeks of registration) of the brain confirming stable CNS disease. Patients with known CNS carcinomatosis or leptomeningeal spread of their disease will be excluded from this study due to their poor prognosis.
4. Patients with gastrointestinal abnormalities including inability to take oral medications, requirement for intravenous alimentation, and malabsorption syndromes will be excluded.
5. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Patients with type I insulin-dependent diabetes or poorly-controlled type II insulin-dependent diabetes or a fasting blood glucose of more than 10 mmol/L (200 mg/dL) will be excluded due to difficulty evaluating the tumor metabolic activity using FDG-PET.
8. History of myocardial infarction or hospitalization for congestive heart failure within 12 months of enrollment.
9. History of prior malignancy (except basal cell carcinoma resected with curative intent) unless resected or treated with curative intent, and disease free for greater than or equal to 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To assess the objective response rate of Panzem NCD alone and in combination with Sunitinib Malate | Throughout study participation

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Liu, MD, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Bruce JY, Eickhoff J, Pili R, Logan T, Carducci M, Arnott J, Treston A, Wilding G, Liu G. A phase II study of 2-methoxyestradiol nanocrystal colloidal dispersion alone and in combination with sunitinib malate in patients with metastatic renal cell carcinoma progressing on sunitinib malate. Invest New Drugs. 2012 Apr;30(2):794-802. doi: 10.1007/s10637-010-9618-9. Epub 2010 Dec 22. PMID 21174224